CLINICAL TRIAL: NCT00084552
Title: Outcomes Following Intensity Modulated Radiation Therapy With And Without Erectile Tissue Dose Sparing For Favorable To Intermediate Risk Prostate Cancer
Brief Title: Intensity-Modulated Radiation Therapy With or Without Decreased Radiation Dose to Erectile Tissue in Treating Patients With Stage II Prostate Cancer
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Fox Chase Cancer Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 03-028; CDR0000365458
Record Dates: First submitted 2004-06-10; First posted 2004-06-11 (Estimated); Results first posted 2021-02-25 (Actual); Last update posted 2021-02-25 (Actual); Status verified 2021-02

CONDITIONS: Prostate Cancer; Sexual Dysfunction; Sexuality and Reproductive Issues
Keywords: sexual dysfunction; sexuality and reproductive issues; adenocarcinoma of the prostate; stage IIB prostate cancer; stage IIA prostate cancer
MeSH Terms: conditions — Prostatic Neoplasms; Sexual Dysfunction, Physiological; Sexuality | interventions — Radiotherapy

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- Arm I (Active Comparator): Patients undergo conventional intensity-modulated radiotherapy (IMRT) once daily 5 days a week for approximately 7.5 weeks.
  Interventions: Radiation: radiation therapy
- Arm II (Experimental): Patients undergo IMRT with dose restriction to erectile tissue once daily 5 days a week for approximately 7.5 weeks.
  Interventions: Radiation: radiation therapy

INTERVENTIONS:
Radiation: radiation therapy — Patients undergo conventional intensity-modulated radiotherapy (IMRT) once daily 5 days a week for approximately 7.5 weeks.

SUMMARY:
RATIONALE: Radiation therapy uses high-energy x-rays to damage tumor cells. Intensity-modulated radiation therapy (radiation directed at the tumor more precisely than in standard radiation therapy) may reduce damage to healthy tissue near the tumor. It is not yet known whether reducing the dose of radiation to erectile tissue will help prevent erectile dysfunction.

PURPOSE: This randomized phase III trial is studying intensity-modulated radiation therapy alone to see how well it works compared to intensity-modulated radiation therapy with reduced doses to erectile tissue in treating patients with stage II prostate cancer.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* Compare erectile dysfunction in patients with stage T1b-T2c adenocarcinoma of the prostate after treatment with intensity-modulated radiotherapy with vs without dose sparing for erectile tissue.

Secondary

* Compare biochemical freedom from failure rates, as a measure of prostate cancer control, in patients treated with these regimens.
* Compare the quality of life of patients treated with these regimens.
* Determine the association of molecular markers and biochemical freedom from failure rate and other endpoints in patients treated with these regimens.

OUTLINE: This is a randomized, single-blind study. Patients are stratified according to age (≤ 65 vs > 65), prescription radiotherapy dose (74 Gy vs 76 Gy), and frequency of erection during sexual activity within the past 4 weeks (a few times vs sometimes vs most times to always). Patients are randomized to 1 of 2 treatment arms.

* Arm I: Patients undergo conventional intensity-modulated radiotherapy (IMRT) once daily 5 days a week for approximately 7.5 weeks.
* Arm II: Patients undergo IMRT with dose restriction to erectile tissue once daily 5 days a week for approximately 7.5 weeks.

Treatment in both arms continues in the absence of unacceptable toxicity or disease metastasis.

Quality of life is assessed at baseline, at 6 and 12 months, and then annually for 4 years

Patients are followed at 3 months and then every 6 months thereafter.

PROJECTED ACCRUAL: A total of 200 patients (100 per treatment arm) will be accrued for this study within 2.5 years.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically confirmed adenocarcinoma of the prostate

  * Clinical stage T1b-T2c by palpation
* Pretreatment prostate-specific antigen ≤ 20 ng/mL
* Gleason score ≤ 7
* Suitable erectile function, defined as a response ≥ score 2 in question #1 of the International Index of Erectile Function Questionnaire
* No clinical, radiographic, or pathologic evidence of nodal or distant metastatic disease

PATIENT CHARACTERISTICS:

Age

* Not specified

Performance status

* Zubrod 0-1

Life expectancy

* Not specified

Hematopoietic

* Not specified

Hepatic

* Not specified

Renal

* Not specified

Other

* Fertile patients must use effective contraception
* No other active malignancy within the past 5 years except nonmetastatic skin cancer or early-stage chronic lymphocytic leukemia (well-differentiated small cell lymphocytic lymphoma)
* No other medical condition that would preclude study participation

PRIOR CONCURRENT THERAPY:

Biologic therapy

* Not specified

Chemotherapy

* Not specified

Endocrine therapy

* Prior androgen-ablation therapy allowed provided total calculated duration ≤ 4 months

Radiotherapy

* No prior pelvic radiotherapy

Surgery

* No prior or planned radical prostate surgery

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 116 (Actual)
Dates: Start 2003-12-11 (Actual); Primary Completion 2013-08-24 (Actual); Study Completion 2016-05-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Eric Horwitz, MD, Principal Investigator — Fox Chase Cancer Center
Locations (1):
- Fox Chase Cancer Center - Philadelphia, Philadelphia, Pennsylvania, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- Standard IMRT (S-IMRT): Patients undergo conventional intensity-modulated radiotherapy (IMRT) once daily 5 days a week for approximately 7.5 weeks.
  radiation therapy: Patients undergo conventional intensity-modulated radiotherapy (IMRT) once daily 5 days a week for approximately 7.5 weeks.
- Erectile Tissue Sparing IMRT (ETS-IMRT): Patients undergo IMRT with dose restriction to erectile tissue once daily 5 days a week for approximately 7.5 weeks.
  radiation therapy: Patients undergo conventional intensity-modulated radiotherapy (IMRT) once daily 5 days a week for approximately 7.5 weeks.
Period: Overall Study
Arm/Group | Standard IMRT (S-IMRT) | Erectile Tissue Sparing IMRT (ETS-IMRT)
Started | 54 | 62
Completed | 54 | 62
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- s-IMRT: Patients undergo conventional intensity-modulated radiotherapy (IMRT) once daily 5 days a week for approximately 7.5 weeks.
  radiation therapy: Patients undergo conventional intensity-modulated radiotherapy (IMRT) once daily 5 days a week for approximately 7.5 weeks.
- ETS-IMRT: Patients undergo IMRT with dose restriction to erectile tissue once daily 5 days a week for approximately 7.5 weeks.
  radiation therapy: Patients undergo conventional intensity-modulated radiotherapy (IMRT) once daily 5 days a week for approximately 7.5 weeks.
- Total: Total of all reporting groups
Arm/Group | s-IMRT | ETS-IMRT | Total
Number analyzed (Participants) | 54 | 62 | 116
Age, Continuous [Median (Full Range); unit: years] | 61 [47 to 75] | 62 [42 to 77] | 62 [42 to 77]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0
  Male | 54 | 62 | 116
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White | 44 | 51 | 95
  Black | 10 | 10 | 20
  Hispanic | 0 | 1 | 1
Region of Enrollment [Number; unit: participants]
  United States | 54 | 62 | 116

OUTCOME MEASURES:

1. Primary Outcome: Erectile Dysfunction Rates
Description: Postage Stamp Test
  -A row of stamps is placed around the base of the penis and the ends are moistened and joined. If the circle is broken in the morning then the subject was recorded as having had a nocturnal erection
  International Index of Erectile Function (IIEF) Questionnaire
  * 15-item questionnaire that measures erectile function
  * Includes companion questionnaire which measures how the partner feels her sexual relationship with the patient has changed since his cancer diagnosis and therapy
Time Frame: 5 year duration after completion of radiotherapy
Population: Some patients did not submit follow-up questionnaires at 24 months post-treatment
Measure: Count of Participants; unit: Participants
Arm/Group | s-IMRT | ETS-IMRT
Number analyzed (Participants) | 37 | 48
Participants | 27 | 36

2. Secondary Outcome: Percentage of Patients With Freedom From Biochemical Failure
Description: Patients without documented failure will undergo needle biopsy of the prostate. A minimum of 12 core biopsies will be taken and additional biopsies will be taken from any suspicious areas (ultrasound or palpation) and/or the original site of biopsy confirmation of prostate cancer at diagnosis. The 12 biopsy sites include sextant, bilateral lateral base, bilateral lateral mid-gland and bilateral transition zone. These data will enable us to evaluate the extent of disease eradication, as well as the prognostic significance of positive biopsies in otherwise palpably normal prostate glands after treatment.
Time Frame: 2 years after treatment
Measure: Number; unit: percentage of participants
Arm/Group | s-IMRT | ETS-IMRT
Number analyzed (Participants) | 54 | 62
percentage of participants | 90.7 | 91.8

3. Secondary Outcome: Acute GI Toxicity
Time Frame: 5 years after treatment
Measure: Count of Participants; unit: Participants
Arm/Group | s-IMRT | ETS-IMRT
Number analyzed (Participants) | 54 | 62
Participants | 1 | 6

4. Secondary Outcome: Acute GU Toxicity
Time Frame: 5 years after treatment
Measure: Count of Participants; unit: Participants
Arm/Group | s-IMRT | ETS-IMRT
Number analyzed (Participants) | 54 | 62
Participants | 20 | 27

ADVERSE EVENTS:
Time Frame: 5 years
Arm/Group | s-IMRT | ETS-IMRT
All-Cause Mortality (participants affected / at risk) | 0/54 | 0/62
Serious Adverse Events (participants affected / at risk) | 0/54 | 0/62
Other Adverse Events (participants affected / at risk) | 0/54 | 0/62

LIMITATIONS AND CAVEATS:
The magnitude of the effect of erectile sparing constraints may be decreased for patients who experience dose-limiting parameters in the s-IMRT arm.

Some patients did not complete follow-up, and to submit follow-up questionnaires at 24 months post-treatment.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes